CLINICAL TRIAL: NCT05370482
Title: Magnetic Resonance Imaging-guided Focal Laser Ablation of Prostate Cancer
Brief Title: MRI-guided Focal Laser Ablation Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13069
Record Dates: First submitted 2022-05-06; First posted 2022-05-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-05

CONDITIONS: Prostate Neoplams, Magnetic Resonance Imaging, Laser Ablation

STUDY DESIGN:
Intervention Model Description: CLS, Tranberg, Laser system
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MRI-guided focal laser ablation (Experimental)
  Interventions: Device: Focal laser ablation

INTERVENTIONS:
Device: Focal laser ablation — MRI-guided focal laser ablation for prostate cancer

SUMMARY:
Prostate cancer is the most frequent malignancy in the male population of developed countries and has a substantial socio-economic impact. Focal therapies, including focal laser ablation (FLA), are gaining ground as a novel strategy to treat organ-confined low- to intermediate risk PCa while preserving healthy tissue and reduce treatment-related morbidity associated with radical treatments.

This project has the goal to perform a feasibility study on magnetic resonance imaging (MRI)-guided focal laser ablation using the TRANBERG®|Thermoguide Therapy System including TRANBERG®Thermoguide Workstation for MR thermometry developed by the company CLS AB.

DETAILED DESCRIPTION:
Prostate cancer is the most frequent non-cutaneous malignancy in the western male population, with almost 13,600 newly diagnosed patients in the Netherlands in 2019. Due to widespread use of the prostate-specific antigen (PSA) test and the lowered PSA threshold for biopsy, the number of newly diagnosed prostate cancers strongly increased in the last 20 years.

At present, treatment choice for prostate cancer patients at low or intermediate risk of disease progression lies between active surveillance (AS) and radical therapies, such as radical prostatectomy or radiotherapy. For these patients, radical treatments have a comparable effectiveness, with a risk of specific death of less than 1% in 15 years. However, none is devised of consequences on the quality of life and can induce significant morbidities such as incontinence and impotence.

For this reason, innovative ablation techniques such as cryosurgery, high intensity focused ultrasound, photodynamic therapy and laser ablation therapy have emerged and are increasingly applied in clinical practice. These treatment methods aim for local destruction of cancerous cells using various sources of energy. The main advantage of preservation of healthy prostatic tissue is to reduce treatment-related complications and morbidity. Recent studies demonstrate that post-treatment prognosis is predominantly driven by the largest lesion with the highest grade, the so-called 'index lesion'. Treatment approaches which preserve parts of the prostatic gland are considered as focal therapy. Imaging plays an important role in detection, localization, targeting and monitoring of focal prostate cancer treatment. Multi-parametric magnetic resonance imaging (mpMRI) is preferred in detecting and staging prostate cancer due to excellent soft tissue contrast and multiplanar anatomical imaging. It is also used to differentiate between post-treatment changes and potential recurrent or residual disease. As such, secondary treatment can be promptly established. More recently, mpMRI has gained acceptance in image-guided therapeutic settings since it offers real-time anatomical imaging in different planes and therefore improved treatment accuracy. Furthermore it can provide real-time temperature imaging.

Focal laser ablation (FLA) or laser-induced interstitial thermal therapy (LITT) is a relatively new technique which was originally developed to treat brain tumors. During this therapy, a laser fiber is positioned into the tumor under image guidance (ultrasound or MRI). When the position of the fiber is correct, laser light is delivered through the fiber and the temperature of the tissue around the tip of the fiber increases. When temperature increases above 60°C the tissue is irreversibly damaged and destroyed. The total ablation process takes about 2-3 minutes. MRI is perfectly suited to use for image guidance during FLA, because it can be used to localize the tumor, target it with probes, monitor and control the ablation procedure in real-time and to map tissue temperature.

Only a few studies on MRI-guided FLA are known. Lepor et al provided a pilot study of 25 patients with low-intermediate risk prostate cancer undergoing FLA. Three months after treatment, they showed no significant differences in functional outcome according to the SHIM (Sexual Health in Man) and AUASS (American Urological Association Symptom Score) questionnaires and no incontinence. Furthermore, 96% of the ablation zones targeted with biopsy three months after treatment, showed no histopathological prove of residual prostate cancer. A recent study by Walser et al. demonstrated a freedom of retreatment rate of 83% after a one year follow up in a group of 120 men with low- to intermediate risk disease that underwent transrectal FLA with no significant changes in quality of life or sexual and urinary function.

In Radboudumc we have several years of experience with MRI-guided focal laser ablation for prostate cancer treatment. At this moment separate systems are used for MR thermometry (IFE, Siemens) and laser energy control (Biolitec). CLS offers a dedicated system which integrates laser energy control with MR thermometry for ablation monitoring. Next to this, additional types of laser fibers are available that are thought to produce relatively larger, more adequate ablation zones (up to 3.0 x 2.0 cm) in comparison to current fibers. In potential, this will decrease the total procedure time because less ablations per lesion are needed and more patients will be eligible for FLA because larger tumors can be treated.

This project has the purpose to assess the feasibility of MRI-guided FLA treatment using the newly developed CLS system as well as its usability and safety.

ELIGIBILITY:
Inclusion Criteria:

* MRI visible index lesion (on T2-weighted MR imaging or diffusion weighted imaging);
* maximum MRI visible lesion size is ≤ 20 mm large axis;
* age 45 to 76 years old;
* life expectancy at inclusion of more 10 years;
* diagnosis of prostate cancer confirmed by targeted biopsy;
* criteria of low and intermediate risk of progression and eligibility for focal therapy;

  * clinical stage of maximum T2c
  * maximum biopsy Gleason score of 4 + 3 on targeted biopsies
  * serum prostate specific antigen < 15 ng/ml
* patient accepting to be included in an active surveillance protocol at the end of the study, in accordance with the recommendations of good practice.

Exclusion Criteria:

* History of prostate surgery;
* history of radiation therapy or pelvic trauma; history of proved acute or chronic prostatitis;
* history of tumor in the preceding 5 years (excluded: non-metastatic basal cell skin cancer);
* severe urinary symptoms associated with benign hyperplasia of the prostate, and defined by an IPSS score > 18;
* tumor with extra-capsular extension or invasion of the seminal vesicles;
* patients with >2 lesions;
* impossibility to obtain a valid informed consent;
* patients unable to undergo MR imaging, including those with contra-indications;
* contra-indications to MR guided focal laser therapy (colitis ulcerosa, rectal pathology or abdomino perineal resection);
* metallic hip implant or any other metallic implant or device that distorts local magnetic field and compromises the quality of MR imaging;
* patients with evidence for nodal or metastatic disease;
* patients with an estimated Glomerular Filtration Ratio (eGFR) < 40 mL/min/1.73 m2

Ages: 45 Years to 76 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-04-11 (Actual); Primary Completion 2023-10-11 (Estimated); Study Completion 2025-04-11 (Estimated)

PRIMARY OUTCOMES:
completion of complete ablation without technical failures | 1 day
  completion of laser ablation without technical failures, achievement of complete ablation shown by MRI after treatment calculated using image co-registration software, total procedure time, total numver of fiber positions and ablations needed
procedure-related adverse events and complications following SIR criteria | 6 months
  procedure-related adverse events and complications following SIR criteria

SECONDARY OUTCOMES:
tumor response | 6 months
  measured with MRI 6 months after treatment
(local) progression free survival (PFS) at 6 months | 6 months
  measured with MRI
incontinence en potency rate | 6 months
  according to IPSS and IIEF-5

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Fütterer, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No